CLINICAL TRIAL: NCT05018884
Title: Incidence, Microbial Spectrum and Risk Factors of Surgical Site Infections at a West Cameroon Hospital: A Prospective Cohort Study
Brief Title: Surgical Site Infections at a West Cameroon Hospital
Acronym: SSI Mbouo
Status: Completed | Type: Observational
Sponsor: Christian Doll (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor-Investigator, Christian Doll, Dr. med. Christian Doll, Universite Evangelique du Cameroun
Organization: Universite Evangelique du Cameroun (Other)
Other Study IDs: SSI Mbouo
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Surgical Wound Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without SSI: Patients who underwent surgery and who developed a surgical site infection (SSI) during 30 days after surgery
- Patients with SSI: Patients who underwent surgery and who didn't develop a surgical site infection (SSI) during 30 days after surgery
  Interventions: Procedure: Observation of surgical site infections

INTERVENTIONS:
Procedure: Observation of surgical site infections — No intervention is done, only observation of routine clinical practice
  Groups: Patients with SSI

SUMMARY:
Surgical site infections (SSI) constitute an important health concern in low and middle income countries, leading to prolonged hospital stay and increased costs. Previous studies indicate that in Africa up to 1/3 of patients undergoing surgery may be affected by a postoperative infection. The development and implementation of context-specific SSI prevention guidelines is important to reduce this complication. To deploy efficient context-specific measures, data on epidemiology and microbiology of these infections are needed. This means to adapt the prevention measures to the context-specific risk factors for surgical site infections in resource-limited settings, and to give locally adapted recommendations on antimicrobial therapy based on local resistance patterns. However, data in this respect are scarce in low and middle income countries. This present study will contribute to the needed epidemiology and microbiology data on SSI in Cameroon. It will be carried out as a prospective cohort study at the Mbouo Protestant hospital in the West Region of Cameroon. The incidence, microbial spectrum and respective antimicrobial resistance of SSI as well as the risk factors of SSI will be systematically investigated. The study will include 300 patients at the Hôpital Protestant de Mbouo (HPM) who underwent surgery and gave their informed consent for inclusion, the timeframe is 04/2021 - 11/2021. An active SSI surveillance system will be put in place for 30 postoperative days to diagnose SSI.

Expected outcomes:

The incidence of SSI is likely to be higher than 10%. Concerning risk factors, preoperative bodywashing and perioperative antibioprophylaxis is expected to be protective against SSI. Up to 1/3 of SSI are expected to occur after hospital discharge. For the microbial spectrum, a high proportion of Staphylococcus aureus is likely to be found. For the antimicrobial resistance no estimation can be give as data is non-existent in that region from the literature.

ELIGIBILITY:
Inclusion Criteria:

* Patient underwent surgery at the hospital during study period

Exclusion Criteria:

* Unconscious patients, mentally ill patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that receive surgery at the Hôpital Protestant de Mbouo in Cameroon and that are willing and consenting to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Surgical Site Infections (SSI) | 04 / 2021 - 11 / 2021
  The incidence of SSI of all patients included in the study

SECONDARY OUTCOMES:
Risk factors of SSI | 04 / 2021 - 11 / 2021
  What are the risk factors for Surgical site infections?
Microbial spectrum of SSI | 04 / 2021 - 11 / 2021
  What is the microbial spectrum of Surgical site infections?
Post-operative mortality | 04 / 2021 - 11 / 2021
  What is the postoperative mortality of all patients included in the study during hospitalisation for a maximum of 30 days after surgery?

CONTACTS AND LOCATIONS:
Overall Officials: Christian Doll, Dr, Principal Investigator — Université Evangélique du Cameroun, Cameroon; Hôpital Protestant de Mbouo, Cameroon; Charité University Medical Centre Berlin, Germany; University Medical Centre Jena, Germany
Locations (1):
- Hôpital Protestant de Mbouo, Bafoussam, West Region, Cameroon

IPD SHARING:
Plan to Share IPD: Undecided
After the end of the study, IPD may be shared on request by other researchers

REFERENCES:
- [Derived] Doll C, Ndoho Simo LC, Jeulefack H, Tamuedjoun Talom A, Kuate Kamdem L, Kenmogne JB, Djeunang Dongho GB, Trampuz A. Efforts in surgical site infection surveillance at the Mbouo Protestant Hospital in Cameroon. BMC Surg. 2025 Oct 3;25(1):419. doi: 10.1186/s12893-025-03229-5. PMID 41044533